CLINICAL TRIAL: NCT06359873
Title: To Investigate the Early Warning Effect of CHA2DS2-VASc Score and Left Atrial Diameter on Atrial Fibrillation in Patients With Hypertension
Brief Title: Left Atrial Enlargement: A Crucial Indicator for Identifying Atrial Fibrillation in Patients With Hypertension
Status: Completed | Type: Observational
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Prof. Yuehui Yin, Director, Head of Cardiovascular Medicine, Principal Investigator, Clinical Professor, The Second Affiliated Hospital of Chongqing Medical University
Other Study IDs: LAD-AF
Record Dates: First submitted 2024-03-26; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation; Hypertension,Essential; Left Atrial Dilatation
MeSH Terms: conditions — Atrial Fibrillation; Essential Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Discovery dataset: The electronic medical records of inpatients with primary hypertension from March 2012 to February 2018 were collected from the electronic medical record system of the Second Affiliated Hospital of Chongqing Medical University, and the data were derived from electronic case reports. To ensure robustness, the investigators applied the createDataPartition function in the caret package to randomly split the dataset into a discovery dataset (70%) and an internal validation dataset (30%).
  Interventions: Diagnostic Test: CHA2DS2-VASc score, C2HEST score, and left atrial diameter (LAD)
- Internal validation dataset: The datasets utilized in this study were sourced from the electronic medical record system of the Second Affiliated Hospital of Chongqing Medical University. The investigators applied the createDataPartition function in the caret package to randomly split the dataset into a discovery dataset (70%) and an internal validation dataset (30%).
  Interventions: Diagnostic Test: CHA2DS2-VASc score, C2HEST score, and left atrial diameter (LAD)
- External validation dataset: The electronic medical record data of patients who came from other hospitals based in Chongqing from October 2011 to November 2021 were extracted from the DEMR database of the Medical Data Institute of Chongqing Medical University as external validation dataset.
  Interventions: Diagnostic Test: CHA2DS2-VASc score, C2HEST score, and left atrial diameter (LAD)

INTERVENTIONS:
Diagnostic Test: CHA2DS2-VASc score, C2HEST score, and left atrial diameter (LAD) — CHA2DS2-VASc Score: Congestive heart failure (HF) [1 point], hypertension [1 point], age ≥ 75 years [2 points], diabetes [1 point], prior stroke or transient ischemic attack [2 points], vascular disease [1 point], age 65-74 years [1 point], and female gender[1 point].
  C2HEST Score: Coronary artery disease or chronic obstructive pulmonary disease [1 point each, 2 total points]; hypertension [1 point]; elderly [2 points for age ≥ 75 years]; systolic HF [2 points]; and thyroid disease [1 point for hyperthyroidism][10].
  LAD: The LAD values of the enrolled patients were extracted by keyword search based on the results of echocardiography in the database.

SUMMARY:
Based on the data of inpatients with hypertension and a cross-sectional study with a large sample size, this study aims to find the early warning value of the left anteroposterior atrial diameter for the possible occurrence of atrial fibrillation in patients with hypertension, and compare the advantages and disadvantages of the above two methods for the early warning of the risk of atrial fibrillation in patients with hypertension, so as to achieve the purpose of early identification of high-risk groups that may develop atrial fibrillation.

DETAILED DESCRIPTION:
Background Left atrial enlargement resulting from hypertension is closely linked to the development and persistence of atrial fibrillation (AF). The newly proposed staging recognizes AF as disease continuum, which makes us aware that AF prevention should focus on the Pre-AF stage, and atrial enlargement is one of the important manifestations in this stage. Previous scoring systems, such as CHA2DS2-VASc and C2HEST, along with the recently highlighted left atrial diameter (LAD), have been significant tools for predicting AF occurrence. However, a comprehensive assessment of their utility is currently lacking.

Purpose This study aims to explore the role of left atrial size in identifying atrial fibrillation (AF) among hospitalized hypertensives, and to compare its recognition effectiveness with previous scoring systems.

Methods The investigators conducted a cross-sectional analysis within hospitalized hypertensives. The discovery, internal and external validation datasets were established. The eXtreme Gradient Boosting (XGBoost) was employed to identify key variables related to AF occurrence, which were ranked based on their importance scores. To gauge the predictive prowess of LAD regarding AF occurrence, the investigators plotted the receiver operating characteristic curve (ROC) and calculated the area under the curve (AUC). This enabled us to pinpoint the LAD cutoff value corresponding to the maximum Youden index, indicative of susceptibility to AF. Subsequently, Youden index determined the optimal cutoff value from the ROC curve. Delong's test compared the identification abilities of different tools within the same dataset. Logistic regression analysis assessed the correlation between clinical variables and left atrial size.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of primary hypertension using the current or past medical history.
* Availability of one or more complete ECG and 24h holter data.
* Availability of complete echocardiogram data in the current hospitalization.

Exclusion Criteria:

* Patients under 18 years of age.
* Cases with incomplete or unidentifiable results from extracted data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The electronic medical records of inpatients with primary hypertension from March 2012 to February 2018 were collected from the electronic medical record system of the Second Affiliated Hospital of Chongqing Medical University, and the data were derived from electronic case reports. Furthermore, the electronic medical record data of patients in other hospitals from October 2011 to November 2021 were extracted from the DEMR database as external data. The extraction of discharge diagnoses relied on International Classification of Diseases (ICD) hospitalization discharge codes. Patient information within the database was kept anonymous and safeguarded by unique identification numbers to ensure strict confidentiality. Importantly, the retrospective nature of this study had no influence on the medical care processes of the subjects, and it received ethical approval from the Medical Ethics Committee of the Second Affiliated Hospital of Chongqing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 58427 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
left atrial diameter (LAD) | Data collection was completed after discharge from the hospital, up to 3 months.
  In this study, after the patients completed the cardiac color Doppler ultrasound, the report and results would be uploaded to the electronic medical record system. Then, the investigator would extract the LAD values recorded in the report from this database.
CHA2DS2-VASc score | Data collection was completed after discharge from the hospital, up to 3 months.
  The patients' discharge material were extracted from the database, including age, gender, and history of congestive heart failure, hypertension, diabetes, stroke or transient ischemic attacks, and vascular disease. CHA2DS2-VASc score was calculated according to the guidelines (CHA2DS2-VASc criteria: Congestive heart failure [1 point], hypertension [1 point], age ≥ 75 years [2 points], diabetes [1 point], prior stroke or transient ischemic attack [2 points], vascular disease [1 point], age 65-74 years [1 point], and female gender[1 point]), with the highest score being 9 and the lowest score being 0. Then, the CHA2DS2-VASc score was calculated by the investigator based on the above diagnosis. The higher the score, the higher the risk of AF.
C2HEST score | Data collection was completed after discharge from the hospital, up to 3 months.
  The patients' discharge material were extracted from the database, including age, and history of coronary artery disease, chronic obstructive pulmonary disease, hypertension, systolic heart failure, thyroid disease. C2HEST score was calculated according to the guidelines (C2HEST criteria: Coronary artery disease or chronic obstructive pulmonary disease [1 point each, 2 total points]; hypertension [1 point]; elderly [2 points for age ≥ 75 years]; systolic heart failure [2 points]; and thyroid disease [1 point for hyperthyroidism]), with the highest score being 8 and the lowest score being 0. Then, the C2HEST score was calculated by the investigator based on the above diagnosis. The higher the score, the higher the risk of AF.
Atrial fibrillation (AF) | Data collection was completed after discharge from the hospital, up to 3 months.
  Diagnostic criteria for AF: The preferred indicators for confirming the diagnosis of AF were normal ECG and ambulatory ECG. During physical examination, the patient's heart rhythm is absolutely irregular and the first heart sound is uneven in strength. Patients may also present with clinical manifestations such as palpitations, dizziness, dyspnea, and chest tightness during the course of the disease. The above materials of the patients were recorded in the electronic medical record system.

SECONDARY OUTCOMES:
Area under the curve (AUC) of LAD and occurrence of AF | Statistics were completed after data collection, up to 1 months.
  To assess the ability of LAD to predict the occurrence of AF, the investigators used IBM SPSS 26.0 software to create a receiver operating characteristic curve (ROC) and calculate the AUC in the discovery and external datasets, with LAD as the independent variable and the occurrence of AF as the dependent variable.
AUC of CHA2DS2-VASc score and occurrence of AF | Statistics were completed after data collection, up to 1 months.
  To gauge the predictive prowess of CHA2DS2-VASc scores regarding AF occurrence, a ROC was plotted and the AUC was calculated in the discovery and external datasets, with CHA2DS2-VASc score as the independent variable and the occurrence of AF as the dependent variable.
AUC of C2HEST score and occurrence of AF | Statistics were completed after data collection, up to 1 months.
  To gauge the predictive prowess of C2HEST scores regarding AF occurrence, a ROC was plotted and the AUC was calculated in the discovery and external datasets, with C2HEST score as the independent variable and the occurrence of AF as the dependent variable.

OTHER OUTCOMES:
the LAD cutoff value | Statistics were completed after data collection, up to 1 months.
  To facilitate clinical use, as well as to assess the predictive power of LAD for the occurrence of AF, AUC was calculated in the discovery and external datasets. This enabled us to pinpoint the LAD cutoff value corresponding to the maximum Youden index, indicative of susceptibility to AF.

CONTACTS AND LOCATIONS:
Overall Officials: Yuehui Yin, MD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- 2ndChongqingMU, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified electronic medical record (DEMR) data platform of Chongqing Medical University Medical Data Institute, accessible at https://demo.yiducloud.com.cn/pub/#/register.
Supporting Information: CSR
Access Criteria: Researchers need to complete the registration information online, and they can access it after being reviewed by the Institute of Medical Data of Chongqing Medical University.
URL: http://demo.yiducloud.com.cn/pub/#/register.